CLINICAL TRIAL: NCT03668210
Title: Risk Factor of Anterior Cruciate Ligament Rupture After Ligamentoplasty : What is the Importance of a Relative Deficit of Contralateral Hamstrings Assessed by Isokinetic in Postoperative ?
Acronym: DIS-RRACT
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3074
Record Dates: First submitted 2018-09-05; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Anterior cruciate ligament; ligamentoplasty; isokinetics
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with contralateral ACL after Ligamentoplasty: Athletic patients who have consulted in Sports Medicine Department at the Rennes University Hospital, victims of an ACL rupture during sports activity and who declared a contralateral ACL after the ligamentoplasty.
  Isokinetic evaluation.
  Interventions: Procedure: Isokinetic evaluation
- Patients without contralateral ACL rupture: Athletic patients who have consulted in Sports Medicine Department at Rennes University Hospital, without ACL rupture.
  Isokinetic evaluation.
  Interventions: Procedure: Isokinetic evaluation

INTERVENTIONS:
Procedure: Isokinetic evaluation — Isokinetics is used to measure the peak of strength of quadriceps and hamstrings, in concentric or eccentric, at slow and fast speed to determine a hamstring / quadriceps ratio to highlight a deficit or imbalance.

SUMMARY:
Anterior cruciate ligament (ACL) is a common pathology (37 000 operations in 2006, nearly 43 000 in 2012 in France) justifying more and more operating indications in younger and younger patients. 70-80% of ACL ruptures occur without contact, which makes it a major public health interest because of its frequency and accessibility in terms of prevention.

The place of isokinetic assessment is important pre and postoperatively so that it has become systematic.

DETAILED DESCRIPTION:
The main risk factors for known ACL lesions are female gender, pivotal sports, neuromuscular deficits, proprioceptive, hormonal, morphological deficits ... Moreover, there is also an increase in the number of contralateral fractures in patients who had a ligamentoplasty. There are many articles on the ACL pathology but unequal on the potential risk factors. The only proven risk factor for contralateral rupture is the age of the first episode; the female sex also seems to be important in some studies but remains more controversial. However, many factors have been studied: the intensity of the sport, the sex, the operative technique of ligamentoplasty, the operating duration, the duration of recovery of the sports activity, the level of recovery (of this sporting activity ) ...

Isokinetics is used to measure the peak of strength of quadriceps and hamstrings, in concentric or eccentric, at slow and fast speed and to determine a hamstring / quadriceps ratio to highlight a deficit or imbalance.

ELIGIBILITY:
Inclusion Criteria:

* Athletic patients all levels
* victims of ACL rupture during sports practice,
* operated by the same surgeon
* having been evaluated in isokinetic postoperative in the Sports Medicine Department of Rennes University Hospital
* having resumed a sporting activity
* with the first ACL rupture between 01/01/1994 and 12/31/2015

Exclusion Criteria:

* Patients with ACL rupture outside of a sporting context
* not having resumed post-operative sports activity on the maximum follow-up period of 15 years
* not evaluated for isokinetic activity in the sports medicine department
* minors at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Athletic patients who have consulted in Sports Medicine Department at Rennes University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of relative hamstrings deficiency versus quadriceps expressed by a concentric hamstrings/quadriceps ratio | At inclusion
  Isokineticism makes it possible to measure the peak of force of quadriceps and hamstrings. Concentric hamstrings/quadriceps ratio in isokinetic is calculated to detect a relative deficiency if it is below threshold values of 55% at 60 °/s slow speed, or 65% at 180 °/s fast speed.

SECONDARY OUTCOMES:
Investigating whether a lack of recruitment of hamstring at fast speed is a potential risk factor for ACL rupture, by evaluating hamstrings/quadriceps ratio in isokinetics. | At inclusion
  The lack of recruitment of the hamstrings when increasing speed is defined as normal ratios of peaks of force at the two speeds in isokinetic, but with an increase of the ratio hamstrings/Quadriceps in concentric at fast speed lower than 10%, with reference to the value of the ratio hamstrings/Quadriceps at slow speed.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline JAN, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: No